CLINICAL TRIAL: NCT06107478
Title: Parental Perception of Their Child's Emotional Quality of Life in Paediatric Oncology: Pre-post "Magic Massages" Study
Brief Title: Parental Perception of Their Child's Emotional Quality of Life in Paediatric Oncology Before and After "Magic Massages"
Acronym: MASSAYA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Leon Berard (Other)
Collaborators: Institut d'Hématologie et d'Oncologie Pédiatrique (Unknown); Fondation La Roche Posay (Unknown)
Responsible Party: Sponsor
Other Study IDs: ET23000304
Record Dates: First submitted 2023-09-27; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
Keywords: Oncopeadiatrics; Quality of life; Anxiety; Depression; Parental perception; Parent-child-caregiver relationship; Massages
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anxiety Disorders; Depression | interventions — Single Person; Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children ALL, 2-12 years old: Children with acute lymphoblastic leukemia (ALL) and in the induction phase of its treatment (at least one month post-diagnosis and up to 50 days post-diagnosis, i.e. until the first day of consolidation).
  Interventions: Other: Clinical data collection (only concerning Children)
- Parents of children ALL: Parents of a patient with acute lymphoblastic leukemia (ALL) being in the induction phase of his treatment (at least one month post-diagnosis and up to 50 days post-diagnosis, i.e. until the first day of consolidation), 2 to 12 years of age at diagnosis and managed by a participating centre.
  Interventions: Other: Self-report questionnaires (only for parents); Other: Interview (only for parents)

INTERVENTIONS:
Other: Self-report questionnaires (only for parents) — Quantitative part (all investigating centers): When they come to the various timepoints (T0, T1, T2), participants will be asked to fill in self-questionnaires, either electronically or on paper. If they are unable to come to the center at T1 and/or T2, they will be offered the option of completing the self-questionnaires online. These can also be sent by e-mail or postal mail and received by the same means if necessary.
  The tools:
  * Quality of life: Pediatric Quality of Life Inventory
  * Anxiety: Edmonton Symptom Assessment System; Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Scale
  * Depression: Edmonton Symptom Assessment System; PROMIS depression scale
  * Parent-child relationship: Ad hoc questionnaire
  * Parent-caregiver relationship: Enabling Practices Scale Socio-demographic data on parents and children, data relating to supportive care will be collected at inclusion. Massage habits will be collected at T1 and T2.
  Groups: Parents of children ALL
Other: Interview (only for parents) — Qualitative part (exclusively at CLB):
  Participants (parents) in the qualitative part of the study will be asked to complete a self-administered questionnaire on socio-demographic data when they come to the center at T0. Clinical data will also be collected at T0. At T1, an interview will be organized with a researcher dedicated to the study. Qualitative interviews will preferably take place face-to-face, although videoconferencing may be used in certain circumstances.
  Groups: Parents of children ALL
Other: Clinical data collection (only concerning Children) — The children's medical data (patients) will be collected in a Case Report Form (CRF; e.g. type of cancer, date of diagnosis, anti-cancer treatments received, symptoms) at T0.
  Groups: Children ALL, 2-12 years old

SUMMARY:
Rationale: In France, 1,850 cases of cancer are diagnosed in children every year (28% of leukaemia). Despite a cure rate of 83% (all cancers combined), treatment remains a major burden. Changes to the body caused by the disease and its treatment can alter their self-image and the way they relate to their bodies. The massage benefits for children have been highlighted, improving their quality of life (QoL) during treatment. The importance of including parents in the paediatric care process in order to strengthen family ties was also highlighted. Recently, the La Roche-Posay Foundation, in conjunction with a group of experts, developed and rolled out a training course called "Magic Massages" (MM), aimed at parents. The Human and Social Sciences Department of the Léon Bérard Center, in collaboration with the Institute of Paediatric Haematology and Oncology, and with the support of the La Roche Posay Foundation, is conducting a longitudinal multicenter observational study, the main aim of which is to assess parental perceptions of the impact of therapeutic massage on their child's emotional QoL. The secondary objectives of this study are to assess parental perception of the impact of therapeutic massage on their child's QoL and emotional distress (i.e. anxiety and depression), as well as on the quality of the parent-child-caregiver relationship.

Method: In this mixed-method study, 181 parents with a child aged 2 to 12 years treated for acute lymphoblastic leukaemia and diagnosed at least one month previously will be recruited; 161 for the quantitative part, and 20 others will be recruited for the qualitative part. Recruitment will take place nationwide in several oncopaediatric centres. Thus, in the quantitative part of the study, parent participants will complete self-reported measures of their child's QoL, anxiety and depression, as well as parent-child and parent-caregiver relationships. Data will be collected before training (T0); 3 weeks (T1) and 6 weeks after MM training (T2). Concerning the qualitative part, semi-directive interviews will be conducted with participants at T1.

Expected results: The implementation of MM would lead to an improvement in QoL, as well as a reduction in anxiety and depression perceived by parents in their child. An increase in the perceived quality of parent-child-caregiver relationships is also expected. In the long term, large-scale deployment of MM could be envisaged, including in other diseases.

DETAILED DESCRIPTION:
Study Type:

Human and social sciences research (NRIPH), observational, mixed (i.e., quantitative and qualitative), longitudinal and multicenter. The study will involve three measurement phases:

T0: before training in "Magic Massages" (MM) T1: 3 weeks after MM training T2: 6 weeks after MM training

Principal aim:

To describe and compare parental perception of the quality of life/psychosocial health of their child with acute lymphoblastic leukaemia (ALL) before MM training (T0) and 3 weeks after MM training (T1).

Secondary aims:

1. To describe parental perception of the quality of life of their child with ALL before MM training (T0), 3 weeks after MM training (T1) and 6 weeks after MM training (T2).
2. To describe parental perception of emotional distress (anxiety/depression) in their child with ALL before MM training (T0), then 3 weeks (T1) and 6 weeks after MM training (T2).
3. Describe parental perception of the relationship with their child before MM training (T0), then 3 weeks (T1) and 6 weeks after MM training (T2).
4. Describe parental perception of their relationship with the caregiver before MM training (T0), then 3 weeks (T1) and 6 weeks after MM training (T2).
5. Qualitatively collect parents' perceptions of their child's overall quality of life, their relationship with their child and the dynamic established with the healthcare team 3 weeks after MM training (T1).

Study Population:

The study will be systematically offered to all parents of a child with ALL who meet the inclusion criteria, at the time of their visit to an investigating center for any treatment, and who have not yet completed the MM training course.

As the child's (patient's) clinical data will be collected, he or she will also be considered a participant.

Study conduct:

The study will be systematically proposed via the team in charge to all parents of a sick child who meet the inclusion and non-inclusion criteria.

The proposal to participate will be made during the induction phase of the patient's treatment, at the investigating center. At this point, participants will be provided with an information leaflet tailored to the type of study (quantitative or qualitative) and the participant's status (parent or child). A reasonable period of reflection will be allowed.

* At the Centre Léon Bérard, participants will be offered either the qualitative study or the quantitative study. Participants in the qualitative part must not have taken part in the quantitative part, in order to avoid bias due to contamination of responses between the two parts.
* In the other investigating centers, the quantitative study will be offered exclusively to all potential participants.

After obtaining the participants' non-opposition, the study team will schedule the MM training session for the first day of the patient's first phase of treatment consolidation (D1).

In all centers, parents will be trained in MM by a member of the investigating center's healthcare team. This training will be given on a one-to-one basis and will last approximately 30 minutes. The trainer will show the parents how to use the MM kit with their child, which they will be able to take home after the training.

Quantitative part (all investigating centers):

When they come to the various measurement points (T0, T1 and T2), participants (parents) will be asked to fill in self-questionnaires, either electronically or on paper. If they are unable to come to the center at T1 and/or T2, they will be offered the option of completing the self-questionnaires online. These can also be sent by e-mail or postal mail and received by the same means if necessary.

Clinical data will be collected at T0.

Qualitative part (exclusively at CLB):

Participants (parents) in the qualitative part of the study will be asked to complete a self-administered questionnaire on socio-demographic data when they come to the center at T0. Clinical data will also be collected at T0. At T1, an interview will be organized with a researcher dedicated to the study. Qualitative interviews will preferably take place face-to-face, although videoconferencing may be used in certain circumstances.

Expected results:

The use of MM is thought to lead to an improvement in quality of life, as well as a reduction in anxiety and depression perceived by parents in their sick child. An increase in the quality of the parent-child-caregiver relationship is also expected.

ELIGIBILITY:
Criteria for including parents :

* Be the parent of a patient with acute lymphoblastic leukaemia (ALL) in the induction phase of treatment (at least one-month post-diagnosis and up to 50 days post-diagnosis, according to the ALL Together 2023 treatment protocol), aged between 2 and 12 years at diagnosis and under the care of a study investigating center.
* Have agreed to undergo training in the Magic Massage technique at the time of the study and at one of the study's investigating centers
* Be able to understand, speak, read and write French
* Have been informed of the study and not to have objected

Criteria for not including parents:

* Have refused to take part in the "Magic Massages" training during the study or have already done so prior to inclusion.
* Have refused or to be incapable of making an informed objection
* Be the 2nd parent of a patient with ALL for whom a 1er parent is already included in the study.
* Be deprived of liberty by a court or administrative order

Inclusion criteria for children

* Have ALL and be in the induction phase of treatment (at least one-month post-diagnosis and up to 50 days post-diagnosis, according to the ALL Together 2023 treatment protocol).
* Be 2 to 12 years of age at diagnosis
* Be under the care of one of the study's investigating centers
* Have been informed of the study in a manner appropriate to their abilities and not to have opposed it

Criteria for non-inclusion of children:

* Not be followed for the duration of the study
* Have refused to take part in the study
* Be deprived of liberty by a court or administrative order

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be systematically offered to all parents of a child with ALL who meet the inclusion criteria, at the time of their visit to an investigating center for any treatment, and who have not yet completed the magic massages (MM) training course.
  As the child's (patient's) clinical data will be collected, he or she will also be considered a participant.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Psychosocial health quality of life score at T0 and T1 | Timepoint 0 (T0) and Timepoint 1 (T1)
  The emotional quality of life score will be calculated based on the psychosocial health dimension of PedsQL (Pediatric Quality of Life Inventory; 5 items).

SECONDARY OUTCOMES:
Scores for different quality of life dimensions at T0, T1 and T2 | Timepoint 0 (T0), Timepoint 1 (T1) and Timepoint 2 (T2)
  The parental perception of the quality of life relative to the health of their child will be measured thanks to the quality of life scores of PedsQL: physical, emotional, social, school, and total score.
Anxiety and depression scores at T0, T1 and T2 | Timepoint 0 (T0), Timepoint 1 (T1) and Timepoint 2 (T2)
  The parental perception of the emotional distress (anxiety and depression) of the child will be measured through the scores of anxiety and depression, from the PROMIS self-questionnaires and a numerical scale from 0 to 10.
Responses to items concerning the parent-child relationship at T0, T1 and T2 | Timepoint 0 (T0), Timepoint 1 (T1) and Timepoint 2 (T2)
  The parental perception of the relationship with their child will be described on the basis of an ad hoc self-questionnaire built specifically for the MASSAYA study.
Parent/caregiver relationship score at T0, T1 and T2 | Timepoint 0 (T0), Timepoint 1 (T1) and Timepoint 2 (T2)
  Parental perception of the relationship with the caregiver will be measured using a score from the EPS7 self-questionnaire.
Qualitative collection of parents' perceptions of their child's overall quality of life, their relationship with their child and with the healthcare team at T1 | Timepoint 1 (T1)
  The parental perception of the overall QoL of their child and the parent-child-caregiver relationships will be collected qualitatively and described through a semi-directive interview at T1.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique CHRISTOPHE, PR, Study Director — Centre Leon Berard; Amélie ANOTA, PHD, Study Director — Centre Leon Berard

IPD SHARING:
Plan to Share IPD: No